CLINICAL TRIAL: NCT03808350
Title: Stress and Engagement Surrounding ICU Procedures Among Patients, Families and Clinicians
Brief Title: Family Procedural Presence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Intermountain Health Care, Inc. (Other)
Collaborators: University of Utah (Other)
Responsible Party: Principal Investigator, Sarah Beesley, Pulmonologist - Shock Trauma ICU, Intermountain Health Care, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1050086
Record Dates: First submitted 2018-12-26; First posted 2019-01-17 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Patient and Family Engagement

STUDY DESIGN:
Who Masked: Participant
Masking Description: Family members and patients will be told the study is being done to understand engagement, but will not be told about the main intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Families Excluded From Presence at Procedures (Placebo Comparator): Families not invited to remain for ICU procedures
  Interventions: Other: Placebo/Control
- Families Invited to Be Present at Procedures (Active Comparator): Families invited to remain for ICU procedures
  Interventions: Procedure: Families Invited to Be Present at Procedures

INTERVENTIONS:
Procedure: Families Invited to Be Present at Procedures — Family members will be invited (but not required) to remain in the ICU room during procedures, if patients agree
  Arms: Families Invited to Be Present at Procedures
Other: Placebo/Control — Family members will not be invited to remain in the ICU room
  Arms: Families Excluded From Presence at Procedures

SUMMARY:
This study seeks to determine the effect of a quality improvement policy regarding allowing family members to remain in a patient's room during ICU procedures. The investigators hypothesized that our change in policy to invite family members to remain during procedures will improve patient & family engagement and improve long term psychological outcomes after an ICU admission. The study also seeks to determine if inviting family members to remain in a patient's room during ICU procedures will not increase clinician stress.

DETAILED DESCRIPTION:
This is a research study about the effect of a quality improvement policy change regarding family presence at ICU procedures on family and patient engagement, psychological outcomes and stress levels in clinicians. In the study, ICU patients, their family members and ICU clinicians will be surveyed regarding these outcomes, with some surveys obtained prior to a policy change and a second set during a second time period after policy change. The patients and family members will be asked survey questions after the procedure and 3 months later. This study will also evaluate the change in clinician stress related to this policy change, and clinicians will also answer survey questions.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* Able to read & speak English
* Family member of a patient or a patient that has undergone one of these procedures at any point during the ICU stay (if the procedure occurs from Sunday at 8 am to Friday at 12 pm): intubation, central line placement, arterial line placement, bronchoscopy, thoracentesis, chest tube placement, paracentesis and lumbar puncture
* Physician (both attending physicians and trainees) and nurses who work in the ICU during the study period.

Exclusion Criteria:

* Patients for whom no family member can be identified
* Non-English speaking individuals
* Children (<18 years of age)
* Participants with dementia, psychiatric disorder with psychosis, schizophrenia or known cognitive dysfunction (established from chart review, report and/or score greater than or equal to 3 on IQ Code screening).
* Provider who does not want to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-09-14 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Patient & Family Member Engagement | Time of ICU procedure to 48 hours afterwards
  Engagement, as measured by the collaboRATE survey, administered to patients & family members within 48 hours after a procedure in the ICU

SECONDARY OUTCOMES:
Patient & Family Member Stress | Time of ICU procedure to 48 hours afterwards
  Perceived stress of patient & family members, assessed within 48 hours after a procedure in the ICU by the Perceived Stress Scale-4 (PSS-4), measured on a scale from 0 to 16 with high numbers indicating increased level of perceived stress.
Clinician Stress | Time of ICU procedure to 48 hours afterwards
  Clinician stress, as assessed within 48 hours after a procedure in ICU by the visual analog scale, measured on a scale from 1-100 with 100 indicating higher levels of clinician stress.
Procedural Complication Rate | Through 7 days after the ICU procedure
  Complications associated with procedures, including infections associated with central lines
Trainee Satisfaction with Procedure Education | Time of ICU procedure to 24 hours afterwards
  Satisfaction with the education experience among trainees performing procedures, as assessed within 24 hours by a Likert scale from 1-5 with 5 indicating increased satisfaction with education experience and 1 indicating dissatisfaction with education experience.
Patient & Family Member Anxiety & Depression | 3 months after ICU procedure
  Anxiety and depression for patients & family members, assessed at 3 months after the ICU procedure by the Hospital Anxiety and Depression Scale (HADS), measured from 0 to 42 with higher scores indicating more likelihood of anxiety or depression.
Patient & Family Member PTSD | 3 months after ICU procedure
  PTSD for patients & family members, assessed at 3 months after the ICU procedure by the Impact of Event Scale Revised (IES-R), measured from 4 to 88 with a score over 33 indicating likely presence of PTSD.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah J Beesley, MD, Principal Investigator — Intermountain Health Care, Inc.
Locations (1):
- Intermountain Medical Center, Murray, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided
Completely deidentified data may potentially be available to other researchers upon request